CLINICAL TRIAL: NCT00955929
Title: A Randomized Trial of Pharmacological Penile Rehabilitation in the Preservation of Erectile Function Following Bilateral Nerve-Sparing Radical Prostatectomy
Brief Title: Pharmacological Penile Rehabilitation in the Preservation of Erectile Function Following Bilateral Nerve-Sparing Radical Prostatectomy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was interrupted because of failure to recruit the target study population in a reasonable timeframe.
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 09-005
Record Dates: First submitted 2009-08-07; First posted 2009-08-10 (Estimated); Results first posted 2021-11-08 (Actual); Last update posted 2021-11-10 (Actual); Status verified 2021-11

CONDITIONS: Penile Cancer; Erectile Dysfunction; Radical Prostatectomy
Keywords: Penis; PLACEBO; SILDENAFIL CITRATE; TRIMIX; Bimix; Viagra; 09-005; Erectile Dysfunction following Bilateral Nerve-Sparing
MeSH Terms: conditions — Penile Neoplasms; Erectile Dysfunction | interventions — Sildenafil Citrate; Surveys and Questionnaires; Alprostadil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- PRN Sildenafil (Experimental): Placebo QHS (blinded) and sildenafil 100mgs (open-label) as required for sexual relations. The placebo will be omitted on nights that 100mgs is used. Placebo will start within 24-48 hours post-surgery.
  Interventions: Drug: Placebo QHS and sildenafil and questionnaires
- Nightly Sildenafil Arm (Experimental): Patients will be instructed to take sildenafil 50 mg QHS (blinded) except on nights that they are interested in sexual relations, they will then be instructed to use sildenafil 100mgs (open-label) and skip the 50mg dose. Sildenafil treatment will start within 24-48 hours post-surgery.
  Interventions: Drug: Sildenafil and questionnaire
- Combination Therapy Arm (Experimental): Trimix combination (Papavarine 30mg/mL Phentholamine 1mg/mL Prostaglandin E1 10 mcg/mL), at initial dose of 5 units (0.05ml) will be given; the first 2 injections will be done in the MSKCC urology outpatient clinic (if needed, the investigator can determine appropriate amount of injections for patient training).
  Interventions: Drug: Trimix combination (Papavarine 30mg/mL Phentholamine 1mg/mL Prostaglandin E1 10 mcg/mmL) and questionnaires

INTERVENTIONS:
Drug: Placebo QHS and sildenafil and questionnaires — Pts will be offered sildenafil 100 mg to be used before intercourse on an as-required basis. They will be given six 100 mg doses, per month, for a 12-month duration. Each patient in this group will use a placebo pill (blinded) each night, except on a nights that 100mg is taken for the purpose of sexual relations. Patients will be evaluated in the clinic and will complete the questionnaires at baseline (pre-treatment evaluation), 3, 6, 9, 12, 18 and 24 months after the operation. At 12 months postoperatively, all patients will stop treatment. Visits 3, 6, 9, 12, 18, and 24 months will have ±2 week window.
  Arms: PRN Sildenafil
Drug: Sildenafil and questionnaire — Patients will be instructed to take sildenafil 50 mg QHS (blinded) except on nights that they are interested in sexual relations, they will then be instructed to use sildenafil 100mgs (open-label) and skip the 50mg dose. Sildenafil treatment will start within 24-48 hours post-surgery. Patients will be evaluated in the clinic and will complete the questionnaires at baseline (pre-treatment evaluation), 3, 6, 9, 12, 18 and 24 months after the operation. At 12 months postoperatively, all patients will stop treatment. Visits 3, 6, 9, 12, 18, and 24 months will have ±2 week window
  Arms: Nightly Sildenafil Arm
Drug: Trimix combination (Papavarine 30mg/mL Phentholamine 1mg/mL Prostaglandin E1 10 mcg/mmL) and questionnaires — Intracavernous injections of a trimix combination (Papaverine 30mg/mL Phentholamine 1mg/mL Prostaglandin E1 10 mcg/mL) will be injected three times a week, and sildenafil 50mg taken on the other four (non-injection) nights. Injection therapy can be used for the purpose of sexual relations. Patients will be evaluated in the clinic and will complete the questionnaires at baseline (pre-treatment evaluation), 3, 6, 9, 12, 18 and 24 months after the operation. At 12 months postoperatively, all patients will stop treatment. Visits 3, 6, 9, 12, 18, and 24 months will have ±2 week window.
  Arms: Combination Therapy Arm

SUMMARY:
When a bilateral nerve-sparing radical prostatectomy (RP) is performed, recovery of erectile function (rigid erections) is reported for up to 80% of patients, who are less than 60 years old. Erectile function recovery is also impacted by patient age, erectile function before surgery, and the length of time after surgery.

Current evidence from studies suggests that developing erections is important, however, these studies have been small, and the evidence is not definite. Animal studies suggest that erection medication (Viagra, Levitra, Cialis) may protect erection tissue, even in the absence of erections. However, the correct treatment plan is unknown. For example, how often does a man need to take sildenafil (Viagra®) to protect his erectile function or to maximize his erectile function recovery? Is only using erection medication enough for erectile function recovery? Would penile injections, which almost ensure production of an erection, be better than using sildenafil (Viagra®), or might a combination be even better at helping recovery of erections? These are types of questions this study might answer.

ELIGIBILITY:
Inclusion Criteria:

* Male, must be ≥ 18 years of age, with histologically confirmed prostate adenocarcinoma, that is clinically localized to the prostate gland
* Stable sexual relationship for ≥ 6 months
* Open or laparoscopic bilateral nerve-sparing radical prostatectomy
* Baseline score of ≥ 22 on the International Index of Erectile Function Domain (Appendix A)
* Able to speak, read and write in the English language
* Calculated creatinine clearance using the 4 variable MDRD equation based on serum creatinine, age, race, and gender of > 60 cc/min
* Patient is able to walk up two flights of stairs briskly without chest pain
* Patient needs to have their baseline sitting AND standing blood pressure and pulse done at the time of consent

Exclusion Criteria:

* Preoperative or planned postoperative pelvic radiation therapy
* Preoperative or planned postoperative androgen deprivation
* Presence of Peyronie's disease at baseline
* Presence of a penile prosthesis at baseline
* Resection of one or both nerve bundles at surgery
* Any contraindications to sildenafil:

  * Patient is currently using nitrates;
  * Presence of retinitis pigmentosa;
  * Presence macular degeneration;
  * MI or CVA within 3 months;
  * Patient is currently using MAOI medications
* Patient is currently using penile self injection medication (Trimix, Bimix, or PGE-1)
* Patient requiring sildenafil for penetration
* Use of sildenafil within 30 days of consent

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2009-08-06 (Actual); Primary Completion 2020-12-09 (Actual); Study Completion 2020-12-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Mulhall, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | PRN Sildenafil | Nightly Sildenafil Arm | Combination Therapy Arm
Started | 13 | 30 | 33
Completed | 13 | 30 | 33
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PRN Sildenafil | Nightly Sildenafil Arm | Combination Therapy Arm | Total
Number analyzed (Participants) | 13 | 30 | 33 | 76
Age, Continuous [Mean (Full Range); unit: years] | 59.8 [46 to 70] | 54.4 [39 to 68] | 56.1 [43 to 73] | 56.1 [39 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 13 | 30 | 33 | 76
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 2 | 7 | 4 | 13
  White | 10 | 22 | 24 | 56
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 3 | 4
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 13 | 30 | 33 | 76

OUTCOME MEASURES:

1. Primary Outcome: Difference in the Erectile Function (EF) Domain Score of the International Index of Erectile Function (IIEF) Between the 3 Groups at 24 Months.
Time Frame: 2 years
Population: Data were not collected
Arm/Group | PRN Sildenafil | Nightly Sildenafil Arm | Combination Therapy Arm
Number analyzed (Participants) | 0 | 0 | 0

2. Secondary Outcome: The Time to Return of Spontaneous Functional Erections.
Time Frame: 2 years
Population: Data were not collected
Arm/Group | PRN Sildenafil | Nightly Sildenafil Arm | Combination Therapy Arm
Number analyzed (Participants) | 0 | 0 | 0

3. Secondary Outcome: The Time for Patients to Respond to Oral Erectogenic Therapy.
Time Frame: 2 years
Population: Data were not collected
Arm/Group | PRN Sildenafil | Nightly Sildenafil Arm | Combination Therapy Arm
Number analyzed (Participants) | 0 | 0 | 0

4. Secondary Outcome: The Proportion of Patients Who Have Normalization of Their Erectile Function (Normalization of the EF Domain of the IIEF).
Time Frame: 2 years
Population: Data were not collected
Arm/Group | PRN Sildenafil | Nightly Sildenafil Arm | Combination Therapy Arm
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | PRN Sildenafil | Nightly Sildenafil Arm | Combination Therapy Arm
All-Cause Mortality (participants affected / at risk) | 0/13 | 2/30 | 0/33
Serious Adverse Events (participants affected / at risk) | 0/13 | 1/30 | 2/33
Other Adverse Events (participants affected / at risk) | 0/13 | 0/30 | 0/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PRN Sildenafil (N=13) | Nightly Sildenafil Arm (N=30) | Combination Therapy Arm (N=33)
Wound complication, non-infectious (Injury, poisoning and procedural complications) | 0 | 1 | 0
Infection w/ Gr 3/4 neut, Pelvis NOS (Infections and infestations) | 0 | 0 | 1
Pain - Extremity-limb (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2013-02-12): https://cdn.clinicaltrials.gov/large-docs/29/NCT00955929/Prot_SAP_000.pdf